CLINICAL TRIAL: NCT02606565
Title: Acceptability and Efficacy of Umbilical Cord Cleansing With 4% Chlorhexidine for the Prevention of Newborn Infections in Lira District, Northern Uganda: A Randomised Controlled Trial
Brief Title: Efficacy of Umbilical Cord Cleansing With a Single Application of 4% Chlorhexidine for the Prevention of Newborn Infections in Uganda: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Centre For International Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-118
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Omphalitis; Septicaemia
MeSH Terms: conditions — Toxemia | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm: 4% chlorhexidine (Experimental): Neonates randomized to the chlorhexidine arm will have umbilical stump cleansing with a single application of 4% chlorhexidine solution at birth
  Interventions: Biological: Intervention arm: 4% chlorhexidine
- Control arm: Dry cord care (No Intervention): Neonates randomized to the control arm will receive the current standard of cord care (dry cord care)

INTERVENTIONS:
Biological: Intervention arm: 4% chlorhexidine — See previous description
  Arms: Intervention arm: 4% chlorhexidine

SUMMARY:
Background: Nearly all the yearly 3.3 million neonatal deaths occur in low and middle income countries. Infections, including those affecting the umbilical cord (omphalitis) are a significant factor in approximately a third of these deaths. In fact, the odds of all-cause mortality are 46% higher among infants with umbilical cord infection than those without infection. Five large randomized controlled trials in Asia and Sub-Saharan Africa have examined the effect of multiple applications (for at least 7 days) of 4% chlorhexidine (CHX) on the umbilical cord on omphalitis and neonatal death. These studies show a consitent positive effect of multiple applications on omphalitis but not on neonatal mortality. Whereas there is mounting evidence for the effect of 7 day chlorhexidine application, there is no data from Africa and only one study from Asia that examines the effect of a single application of CHX as soon as possible after birth. In this single Asian study, CHX led to a reduction in the risk of mild-moderate omphalitis and neonatal death. It is important, in an African setting to explore the effect of a single application, which is programmatically much simpler to implement than daily application for 7 days. Therefore, the investigators' study will compare umbilical cord cleansing with a single application of 4% chlorhexidine at birth with dry cord care in both community and facility births on omphalitis and severe illness in the neonatal period.

Methods: The chlorhexidine study is a community based, individually randomised controlled trial conducted on 4,760 mother-infant pairs in Uganda. The primary outcomes are severe illness and umbilical cord infection (omphalitis). Severe illness is defined as any illness associated with at least one of the following danger signs observed by study research assistants: inability to drink or breastfeed or (a history of) convulsions, lethargy or unconsciousness, vomiting of all feeds, and/or results in hospitalization and/or results in death.

Discussion: This study will provide novel evidence, from a Sub-Saharan African setting of the effect of umbilical cord cleansing with a single application of 4% chlorhexidine at birth in both community and facility births.

ELIGIBILITY:
Inclusion Criteria:

* Newborns weighing 1.5kg or more at birth
* Newborns born to mothers whose HIV I status is negative

Exclusion Criteria:

* Newborns with severe congenital anomalies
* Newborns with infection of the umbilical cord at birth
* Twins or triplets
* Severely ill infants requiring hospitalization immediately after birth
* Children of mothers who cannot appropriately give consent within 12 h of birth

Max Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4760 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Proportion of infants with severe illness | First 28 days of life
  Severe illness will be defined as an acute illness that is associated with any of the following danger signs observed or verified by a study clinician: inability to feed or vomiting of everything and unable to keep anything down, lethargy or unconsciousness, severe lower chest in-drawing, axillary temperature of ≥38.0 degrees Celsius or <35.5 degrees Celsius, grunting, cyanosis, convulsions or a history of convulsions, and/or results in hospitalization and/or results in death. Hospitalization and death resulting from violent injury or burns will not contribute to the severe illness definition.
Proportion of infants with omphalitis | First 28 days of life
  This outcome will be recorded as present or absent based on specific signs. These include: pus, redness (inflammation) and swelling (oedema) of the cord stump and the surrounding skin at its base. Swelling and redness will be further broken down into: none, mild, moderate and severe. No swelling or redness will be the absence of visible swelling or redness; mild swelling or redness as that limited to the cord stump only; moderate swelling or redness as that extending less than 2cm onto the abdominal skin at the base of the stump and severe swelling or redness as extending ≥2cm into the abdominal skin at the base of the stump. Pus will be defined as either present or absent. Cord infection will then be defined based on combinations of these recorded signs and their severity into four categories as follows: 1) redness extending to skin or pus, 2) moderate or severe redness, 3) moderate or severe redness with pus, or severe redness alone and 4) Severe redness with pus.

SECONDARY OUTCOMES:
Death | First 28 days of life
Adverse events | First 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Nankabirwa, MD, MPH, PhD, Principal Investigator — Department of Epidemiology and Biostatistics, School of Public Health, College of Health Sciences, Makerere University
Locations (1):
- Health Centers in Mukono and Kampala districts, Kampala, Uganda

REFERENCES:
- [Result] Imdad A, Bautista RM, Senen KA, Uy ME, Mantaring JB 3rd, Bhutta ZA. Umbilical cord antiseptics for preventing sepsis and death among newborns. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD008635. doi: 10.1002/14651858.CD008635.pub2. PMID 23728678
- [Derived] Nankabirwa V, Tylleskar T, Tumuhamye J, Tumwine JK, Ndeezi G, Martines JC, Sommerfelt H. Efficacy of umbilical cord cleansing with a single application of 4% chlorhexidine for the prevention of newborn infections in Uganda: study protocol for a randomized controlled trial. Trials. 2017 Jul 12;18(1):322. doi: 10.1186/s13063-017-2050-0. PMID 28701228